CLINICAL TRIAL: NCT02535039
Title: Methylprednisolone Combined Electric-acupuncture Treatment Effects on Cognitive Function After Surgery for Elderly Patients With General Anesthesia
Brief Title: Methylprednisolone Combined Electric-acupuncture on Cognitive Function
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Yanchao Yang, resident doctor, Shengjing Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Shengjing hospital
Record Dates: First submitted 2015-05-29; First posted 2015-08-28 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-12

CONDITIONS: Postoperative Complication; Cognitive Retention Disorder
Keywords: Elderly; cognitive retention disorder; methylprednisolone
MeSH Terms: conditions — Postoperative Complications; Memory Disorders | interventions — Methylprednisolone; meprednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Before anesthesia induction, with electroacupuncture can cave, inside the closed cavity, foot three mile point, cupping model for continuous wave type, current pulse frequency of 2 hz, adjust the intensity of the electric acupuncture, with patients complained of needle feeling, can accept no pain and discomfort.Intraoperative sustained electroacupuncture.The same volume of physiological saline will be given.
  Interventions: Other: Physiological saline
- Methylprednisolne (Experimental): in the anaesthesia to 1 mg/kg intravenous methylprednisolone, methylprednisolone continuous use 1 mg/kg * d until the third day after surgery.Before anesthesia induction, with electroacupuncture can cave, inside the closed cavity, foot three mile point, cupping model for continuous wave type, current pulse frequency of 2 hz, adjust the intensity of the electric acupuncture, with patients complained of needle feeling, can accept no pain and discomfort.Intraoperative sustained electroacupuncture.
  Interventions: Drug: Methylprednisolone

INTERVENTIONS:
Drug: Methylprednisolone — Anaesthesia in giving 1 mg/kg intravenous methylprednisolone, methylprednisolone (1 mg/kg * d for application to the third day after surgery
  Other Names: meprednisone
  Arms: Methylprednisolne
Other: Physiological saline — The same volume of physiological saline will be given in Placebo group
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
Postoperative cognitive dysfunction (POCD) refers to the patients in the central nervous system complications after general anesthesia and clinical manifestations of mental disorder, anxiety, personality changes, impaired memory, personality, social skills and cognitive function after surgery for this decline is called postoperative cognitive dysfunction.Due to the lack of effective clinical treatments, how to prevent and solve the postoperative cognitive dysfunction has become a difficulty and a focus of research in the field of anesthesia.Methylprednisolone is a new type of cortical hormone, because of its strong anti-inflammatory effect, less adverse reactions, is widely used in clinical anesthesia.Electric acupuncture as a kind of traditional treatments, after years of clinical application and achieved good curative effect in practice.In this paper by comparing brain oxygen saturation, blood biochemical indexes, Montreal cognitive assessment scale (MOCA) on cognitive function in patients with grade indexes, such as observation of methylprednisolone combined electric acupuncture treatment of elderly patients with general anesthesia early after the operation, the influence of cognitive function.

Through comparing the operation of cerebral oxygen saturation, blood biochemical indexes, Montreal cognitive assessment scale (MOCA) on cognitive function in patients with grade indexes, such as observation of methylprednisolone combined electric acupuncture treatment of elderly patients with general anesthesia early after the operation, the influence of cognitive function.

DETAILED DESCRIPTION:
Choose descending colon cancer radical general anesthesia, 80 cases of patients, ASA Ⅱ ~ level III, aged 65 ~ 75, were randomly divided into two groups: anesthesia method selects the tracheal intubation general anesthesia.All Diprifusor propofol used in patients with TCI system, with the initial plasma concentration of 2.0 ug/ml start TCI, and intravenous sufentanil injection 0.15 ug/kg, propofol 1 ug/ml every 1 minute.After the BIS value < 75, start the fentanyl TCI system, maintaining the plasma concentrations of 4 ng/ml, vein to the interaction between rocuronium 0.8 mg/kg, insert the endotracheal intubation after mechanical ventilation.Adjust the propofol infusion control electrical double-frequency index between 45 to 55.The experimental group to give intravenous methylprednisolone 1 mg/kg/sack.And 1 mg/kg * d continuous application to the third day after surgery.

1 day before the surgery, postoperative 1 day, 2 days, 3 days, 7 days the MOCA scale to assess cognitive function after surgery for the patient.(T0) prior to the induction and bi (T1), 24 h after surgery (T2) and 48 h after surgery (T3) extraction in patients with venous blood, adopts the method of enzyme-linked immunosorbent (ELISA) determination of serum IL - 1 beta, IL - 6, Aβ1-42, p- Tau concentration.In rSO2 intraoperative continuous monitoring, and calculate the average rSO2, intraoperative rSO2 down the biggest percentage compared with basic value rSO2 % of Max.And record the occurrence of adverse reactions to special circumstances.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 65 to 75
* The American Society of anesthesiologists (American Society of Anesthesiology, ASA) class Ⅱ ~ III
* With a primary culture of above (including elementary school)
* There is no history of drug allergy.

Exclusion Criteria:

* Central nervous system and history of mental illness
* Taking sedatives or antidepressants history
* Insulin dependent diabetes
* Coronary heart disease
* Cerebral infarction
* Preoperative MOCA score less than 26 points

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Cognitive function evaluation as measured by Montreal cognitive assessment scale score | Cognitive function evaluation 1 day after the surgey

SECONDARY OUTCOMES:
Plasma concentration of IL - 6 | Plasma concentration of IL - 6 1 day after the surgey

OTHER OUTCOMES:
Plasma concentration of IL - 1 | Plasma concentration of IL - 1 1 day after the surgey
Plasma concentration of Aβ1-42 | Plasma concentration of Aβ1-42 1 day after the surgey
Plasma concentration of p - Tau | Plasma concentration of p - Tau 1 day after the surgey

CONTACTS AND LOCATIONS:
Overall Officials: Junchao Zhu, doctor, Study Director — professor
Locations (1):
- Shengjing hospital of China medical university, Shenyang, Liaoning, China